CLINICAL TRIAL: NCT02912416
Title: Efficacy of Probiotics on Iron Status During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProIron 16
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Prevention of Iron Deficiency
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Capsule with probiotics
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Capsule with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Determine the effect of probiotics on improving iron status in a population of healthy, pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, pregnant women, aged 18-42 years, with a singleton gestation
* Inclusion at 10-12 weeks of gestation
* BMI ≥ 18 and ≤ 30 at baseline
* Provide signed and dated informed consent form
* Willing to comply with all study procedures

Exclusion Criteria:

* Serum ferritin level <20 µg/L or Hb<110 g/L at baseline (visit 1)
* Chronic diseases associated with anemia
* Known Thalassemia
* Hyperemesis gravidarum
* Chronic gastrointestinal disease (inflammable bowel diseases; Crohn's disease, Ulcerative Colitis; diarrheal disease)
* Known gluten intolerance, lactose intolerance, milk protein allergy
* Taking antibiotics within four weeks before inclusion
* Blood or plasma donation within three (3) months prior to baseline
* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
* Smoking or use of nicotine-containing products (currently or during the last three [3] months)
* History of alcohol abuse, or excessive intake of alcohol, as judged by the Investigator
* Hypersensitivity to any of the ingredients in the study products
* Any other reason for exclusion, as judged by the Investigator

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Serum ferritin level | Week 28 of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- CuraÖresund, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No